CLINICAL TRIAL: NCT02163356
Title: Phase I Study of Fenretinide (4-HPR, NSC 374551) Lym-X-Sorb (LXS) Oral Powder Plus Ketoconazole Plus Vincristine in Patients With Recurrent or Resistant Neuroblastoma (IND #68,254)
Brief Title: Fenretinide Lym-X-Sorb + Ketoconazole + Vincristine for Recurrent or Resistant Neuroblastoma
Acronym: SPOC2013-001
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: drug supply
Sponsor: South Plains Oncology Consortium (Network)
Collaborators: The Evan Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPOC-2013-001
Record Dates: First submitted 2014-05-27; First posted 2014-06-13 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Recurrent Neuroblastoma; Neuroblastoma
Keywords: neuroblastoma; recurrent; resistant
MeSH Terms: conditions — Neuroblastoma; Recurrence | interventions — Fenretinide; Ketoconazole; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Primary therapy (Experimental): Fenretinide/LXS oral powder 1500 mg/m2/day for 7 days plus ketoconazole 6 mg/kg/day for 7 days plus single dose vincristine (dose escalating) given on day 3. Starting dose of vincristine is 0.75 mg/m2/dose. Followed by 14 days of rest.
  Interventions: Drug: Fenretinide/LXS Oral Powder; Drug: Ketoconazole; Drug: Vincristine

INTERVENTIONS:
Drug: Fenretinide/LXS Oral Powder — Oral Powder
  Other Names: 4-HPR; Fenretinide/Lym-X-Sorb; 4-HPR/LXS
Drug: Ketoconazole — Oral Tablet
  Other Names: Nizoral
Drug: Vincristine — IV
  Other Names: Oncovin; Vincristine Sulfate

SUMMARY:
Currently there is no known effective treatment for recurrent or resistant neuroblastoma. Fenretinide is an anticancer agent that may work differently than standard chemotherapy. It may cause the buildup of wax-like substances in cancer cells called ceramides. In laboratory studies, it was found that if too much ceramide builds up in the neuroblastoma cells, they die.

Fenretinide has been given by mouth as a capsule to many people, including children. When Fenretinide is given in capsules, very little of the drug is absorbed through the intestines into the body. This means patients have to take many capsules of fenretinide by mouth several times a day. In this study, a new oral preparation of fenretinide (called 4-HPR/LXS oral powder) is being tested to see if more fenretinide can be absorbed into the body. 4-HPR/LXS oral powder has been tested previously in a limited number of both children and adult cancer patients.

Ketoconazole, commonly used to treat fungus infections, can increase fenretinide levels in the body by interfering with the body's ability to break down fenretinide. Ketoconazole will be given at the same time as the fenretinide powder.

There is preclinical data that shows that combining fenretinide and vincristine prolonged survival in animal models, therefore, it is hoped that giving the vincristine with fenretinide will work better against the neuroblastoma that either drug given alone.

About 70 children with neuroblastoma have been treated with various versions of the fenretinide powder to date, including about a dozen children that also took the fenretinide powder with ketoconazole, and no toxicities have occurred that limited the dosage and no serious or unexpected side effects occurred. However, vincristine has never been given with fenretinide or fenretinide plus ketoconazole before. Vincristine has been been given before with ketoconazole to both children and adults with neuroblastomas and other cancers.

DETAILED DESCRIPTION:
Fenretinide has been given by mouth as a capsule to many people, including children. When Fenretinide is given in capsules, very little of the drug is absorbed through the intestines into the body. This means patients have to take many capsules of fenretinide by mouth several times a day. In this study, a new oral preparation of fenretinide (called 4-HPR/LXS oral powder) is being tested to see if more fenretinide can be absorbed into the body. 4-HPR/LXS oral powder has been tested previously in a limited number of both children and adult cancer patients.

Ketoconazole, commonly used to treat fungus infections, can increase fenretinide levels in the body by interfering with the body's ability to break down fenretinide. Ketoconazole will be given at the same time as the fenretinide powder.

There is preclinical data that shows that combining fenretinide and vincristine prolonged survival in animal models, therefore, it is hoped that giving the vincristine with fenretinide will work better against the neuroblastoma that either drug given alone.

About 70 children with neuroblastoma have been treated with various versions of the fenretinide powder to date, including about a dozen children that also took the fenretinide powder with ketoconazole, and no toxicities have occurred that limited the dosage and no serious or unexpected side effects occurred. However, vincristine has never been given with fenretinide or fenretinide plus ketoconazole before. Vincristine has been been given before with ketoconazole to both children and adults with neuroblastomas and other cancers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with neuroblastoma either by histological verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines
* Patients must have high-risk neuroblastoma with at least ONE of the following:

  1. Recurrent/progressive disease at any time
  2. Refractory disease (i.e. less than a partial response to frontline therapy)
  3. Persistent disease after at least a partial response to frontline therapy (i.e. patient has had at least a partial response to frontline therapy but still has residual disease by MIBG, CT/MRI, or bone marrow)
* Patients must have at least ONE of the following sites of disease:

  1. Measurable tumor on MRI or CT scan or X-ray
  2. MIBG scan with positive uptake at minimum of one site
  3. Bone marrow with tumor cells seen on routine morphology
* Patients with a history of complete surgical resection of CNS lesions are eligible if there is no evidence of CNS lesions (MRI or CT required) at study entry evaluation and if other entry criteria are met
* Patients must have a performance status of 0, 1 or 2 (Appendix I). Patients who are unable to walk because of paralysis or tumor pain, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have a life expectancy of greater than or equal to 8 weeks
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  1. Must not have received myelosuppressive chemotherapy and/or biologics within 3 weeks of entry onto this study (4 weeks if prior nitrosourea)
  2. Patients must not have received radiation for a minimum of two weeks prior
  3. Patients are eligible 12 weeks after autologous stem cell transplant
  4. Minimum of six weeks is required following prior therapeutic doses of MIBG.
  5. There is no limit on number of prior regimens
  6. Must not have received any hematopoietic growth factors within 7 days/
  7. Prior therapy with fenretinide and/or fenretinide + ketoconazole is allowed if no DLT's were experienced. Prior therapy with other retinoids
* Patients must NOT receive other anti-cancer agents while on study
* Palliative radiation is allowed to sites that will not be used to measure response during this study
* All patients must have adequate organ function defined as:

  1. Hemoglobin greater than or equal to 8.0
  2. ANC greater than or equal to 500 (7 days after last dose of growth factor)
  3. Platelet count: greater than or equal to 50,000 at least one week since last platelet transfusion
  4. Age-adjusted serum creatinine < 1.5 x normal for age
  5. Patient must have normal cardiac function documented by ejection fraction (> 55%) documented by echocardiogram or radionuclide MUGA evaluation or fractional shortening ( > 27%) documented by echocardiogram and EKG must demonstrate no abnormality severe enough to justify cardiac medications and baseline QTc interval less than or equal to 450 msecs
  6. Total bilirubin less than or equal to 1.5 x normal for age
  7. SGPT (ALT) and SGOT (AST) less than or equal to 3 x normal for age
  8. Normal prothrombin time (PT) for age
  9. Baseline hepatitis titers without evidence of acute/active hepatitis
  10. Serum triglycerides < 300mg/dL fasting or on a random plasma test
  11. Serum calcium < 11.6mg/dL
  12. No hematuria and/or proteinuria greater than 1+ on urinalysis
* Patients with a seizure disorder are study eligible if seizures are controlled on anticonvulsants
* Normal lung function as manifested by no dyspnea at rest and no oxygen requirement
* Negative serum beta-HCG in females, and use of effective contraception in males and females of child-bearing potential, is required
* Skin toxicity no greater than grade 1
* Patients with known genetic metabolic conditions, or other ongoing serious medical issues, must be approved by the Study Chair prior to registration

Exclusion Criteria:

* Patients with CNS parenchymal or meningeal-based lesions that are present at study entry evaluation are NOT eligible
* Pregnancy or breast feeding. Due to the potential teratogenic effects of retinoids, pregnant women are NOT eligible. Breast milk feeding by study patient is NOT allowed
* Patients with history of organ and allogeneic stem cell transplantation
* Patients with a known history of allergy to soy products
* Patients with a known history of a severe allergy or sensitivity to wheat gluten
* Patients requiring anti-arrhythmia cardiac medications are NOT eligible
* Prior therapy with fenretinide, or fenretinide + ketoconazole, if DLT's were experienced
* A known history of intolerance to ketoconazole
* A known history of intolerance to vincristine
* Patients on other essential medications for which an interaction with ketoconazole can be expected and for which dose reductions to other essential medications cannot be made in a manner adequate to ensure patient safety
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study
* Active hepatitis
* Baseline cardiac QTc interval > 450 msecs

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | after each subject has completed 1 cycle of therapy (a cycle is 21 days)
  To determine maximum dose of vincristine when given in combination with 4-HPR/LXS and ketoconazole. Subjects will be enrolled in a standard 3 + 3 design and will receive set doses of HPR/LXS and ketoconazole. Vincristine will be escalated with each dose level up to 1.5 mg/m2. If toxicity occurs due to vincristine, the dose level will be expanded or dose decreased to the previous level as appropriate. If toxicity occurs due to ketoconazole, the dose level will be expanded and the ketoconazole dose decreased to 3 mg/kg/day
Side effect profile of drug combination | after each subject receives the drug combination (a cycle is expected to be 21 days)
  The side effect profile of the combination therapy will be compared to known single agent side effects looking for new unique drug interactions.
Assess plasma pharmacokinetics of fenretinide | On day 1 (hour 0, 2, 4, 6), day 7 (hour 0, 2, 4, 6) and day 9 (after 3 pm) for course 1. For courses 2 and 6, day 1 (hour 0, 4 and 6), and day 7 (hour 0, 4, and 6)
  included analysis of metabolites (4-MPR and 4-oxo-HPR) and related plasma sphingolipids

SECONDARY OUTCOMES:
Disease response | every 42 days while on therapy
  within limitations of a phase 1 study. Time frame may be longer if a subject receives more than 6 cycles of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Watt, MD, Study Chair — University of Texas Southwestern Medical Center
Locations (4):
- United States (4):
  - The University of Chicago Medicine Comer Children's, Chicago, Illinois
  - UT Southwestern Medical Center, Dallas, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided